CLINICAL TRIAL: NCT00011024
Title: Prospective Studies of the Use of Self Hypnosis, Acupuncture and Osteopathic Manipulation on Muscle Tension in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000008-01P3 (NIH); P50AT000008-01 (NIH)
Record Dates: First submitted 2001-02-08; First posted 2001-02-09 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Hypnosis; Acupuncture Therapy; Manipulation, Osteopathic

INTERVENTIONS:
Procedure: Self Hypnosis
Procedure: Acupuncture
Procedure: Osteopathic Manipulation

SUMMARY:
We propose to identify patients and families for inclusion in pilot studies of the three modalities. Patients and their families will be asked to participate in these studies.

Our research group has done some preliminary work with the modality of hypnotherapy, but has no experience to date with the other two modalities. The idea to try relaxation techniques was generated by the observation that there is great variation in the degree to spasticity at different times in the same patient with CP. When queried, mothers responded that they were able to get their child to relax and decrease the tension in their muscles by stroking, talking softly, and/or by playing certain types of music. The availability of hypnosis and training in self-hypnosis was presented to several families of our patients. Their understanding and acceptance of this alternate therapy was gratifying. The results of this therapy have been promising and have encouraged us to proceed with this modality and to consider making other nonconventional modalities available to our patients.

We hypothesize that at least one of the two modalities will be accepted readily by patients with CP and their families, and with their acceptance compliance with the method chosen will be at levels of 80 percent or more.

DETAILED DESCRIPTION:
The primary objective of this project is to develop and evaluate two different alternative or complementary medical modalities that have been used in children with cerebral palsy by practitioners in an attempt to decelerate the complications from the neurologic insult and resultant muscle imbalance. The specific aims are: 1) The development and incorporation of two alternative modalities (osteopathic manipulation and acupuncture) into available services in southern Arizona for individuals with cerebral palsy. 2) The evaluation of the uptake of and compliance with the two modalities in the clinical services for cerebral palsy. 3) Conduct pilot studies of each of the two modalities to determine their efficacy in decreasing the degree of muscle tension in children with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of spastic CP who are between 48 months and 21 years of age.
* For the hypnotherapy-control arm the children must have a cognitive level sufficient to allow them to visualize and enter into trance.
* The cognitive level criteria will not apply to the manipulation-acupuncture-control arm of the study.
* No child will be excluded on the basis of gender, race or culture.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-09; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Burris Duncan, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States